CLINICAL TRIAL: NCT00707954
Title: A Clinical Pharmacology Study of Multiple Doses of TA-7284 in Patients With Type 2 Diabetes Mellitus
Brief Title: Safety, Pharmacokinetics and Pharmacodynamics of TA-7284 in Type 2 Diabetic Patients
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Tanabe Pharma Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TA-7284-02
Record Dates: First submitted 2008-06-27; First posted 2008-07-01 (Estimated); Results first posted 2014-04-28 (Estimated); Last update posted 2026-01-08 (Actual); Status verified 2025-12

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Diabetes; TA-7284
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- TA-7284 (Experimental)
  Interventions: Drug: TA-7284
- Placebo of TA-7284 (Placebo Comparator)
  Interventions: Drug: Placebo of TA-7284

INTERVENTIONS:
Drug: TA-7284 — Patients will receive single ascending dose of TA-7284 in each step (4 doses planned: 25, 100, 200 and 400 mg), once daily, 15 days (1 day followed by a 1 day washout period and then 14 consecutive days)
  Arms: TA-7284
Drug: Placebo of TA-7284 — Patients will receive placebo tablets in each step, once daily, 15 days (1 day followed by a 1 day washout period and then 14 consecutive days)
  Arms: Placebo of TA-7284

SUMMARY:
The purpose of this study is to evaluate the safety, pharmacokinetics and pharmacodynamics of TA-7284 orally administered once daily for 15 days (1 day followed by a 1 day washout period and then 14 consecutive days). Dose escalation design is utilized in this study, and dose escalation of TA-7284 will be starting with 25 mg (step 1). Subsequent doses of 100 mg (step 2), 200 mg (step 3) and 400 mg (step 4) are planned after review of the tolerance and PK of the previous step.

ELIGIBILITY:
Inclusion Criteria:

* Clinically stable Type 2 Diabetes Mellitus
* Females without childbearing potential
* Body mass index (BMI) >= 18.5 kg/m2 and <= 39.9 kg/m2
* Hemoglobin A1c levels >= 6.5% and <= 10%
* Fasting blood glucose levels >= 140 mg/dL and <= 270 mg/dL
* Systolic blood pressure >= 95 mmHg and <= 160 mmHg, and diastolic blood pressure >= 50 mmHg and <= 100 mmHg, and pulse rate >= 50 bpm
* Patients who have not been administered anti-diabetic medication within 2 weeks Prior to dosing
* Medicines if necessary for Hypertension or Dyslipidemia should be administered with stable dosage at least 3 months
* Treatment with diet and exercise should be unchanged for more than 3 months

Exclusion Criteria:

* Type 1 Diabetes Mellitus or Secondary Diabetic Mellitus
* History of diabetic complications which need treatment
* Treatment with insulin, thiazolidinediones, thiazide diuretics、beta blockers or systemic steroids within 3 months prior to informed consent
* Serum creatinine > upper limit of the normal range
* Patients with significant complications

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2008-06; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kazuoki Kondo, MD, Study Director — Tanabe Pharma Corporation
Locations (1):
- P-One Clinic, Hachiōji, Tokyo-to, Japan

REFERENCES:
- [Derived] Iijima H, Kifuji T, Maruyama N, Inagaki N. Pharmacokinetics, Pharmacodynamics, and Safety of Canagliflozin in Japanese Patients with Type 2 Diabetes Mellitus. Adv Ther. 2015 Aug;32(8):768-82. doi: 10.1007/s12325-015-0234-0. Epub 2015 Aug 18. PMID 26280756

RESULTS

PARTICIPANT FLOW:
Groups:
- TA-7284 25 mg: TA-7284 25 mg was administered as a single dose, followed by a one-day washout, and multiple doses for 14 days.
- TA-7284 100 mg: TA-7284 100 mg was administered as a single dose, followed by a one-day washout, and multiple doses for 14 days.
- TA-7284 200 mg: TA-7284 200 mg was administered as a single dose, followed by a one-day washout, and multiple doses for 14 days.
- TA-7284 400 mg: TA-7284 400 mg was administered as a single dose, followed by a one-day washout, and multiple doses for 14 days.
- Placebo: Placebo was administered as a single dose, followed by a one-day washout, and multiple doses for 14 days.
Period: Overall Study
Arm/Group | TA-7284 25 mg | TA-7284 100 mg | TA-7284 200 mg | TA-7284 400 mg | Placebo
Started | 12 | 12 | 14 | 13 | 10
Completed | 12 | 12 | 14 | 13 | 9
Not Completed | 0 | 0 | 0 | 0 | 1
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | TA-7284 25 mg | TA-7284 100 mg | TA-7284 200 mg | TA-7284 400 mg | Placebo | Total
Number analyzed (Participants) | 12 | 12 | 14 | 13 | 10 | 61
Age, Continuous [Mean (Standard Deviation); unit: years] | 49 (10.6) | 52.1 (7.6) | 56.2 (8.6) | 56.5 (8.2) | 57.6 (6.3) | 54.3 (8.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 0 | 1 | 4 | 2 | 11
  Male | 8 | 12 | 13 | 9 | 8 | 50

OUTCOME MEASURES:

1. Primary Outcome: Safety: Adverse Events, Adverse Drug Reactions
Description: In the safety analysis population, adverse events incidences and adverse drug reactions incidences were calculated by dose.
Time Frame: 19 days
Measure: Number; unit: percentage of incidences
Arm/Group | TA-7284 25 mg | TA-7284 100 mg | TA-7284 200 mg | TA-7284 400 mg | Placebo
Number analyzed (Participants) | 12 | 12 | 14 | 13 | 10
percentage of incidences
  Adverse events | 75.0 | 66.7 | 35.7 | 46.2 | 80.0
  Adverse drug reactions | 50.0 | 16.7 | 7.1 | 7.7 | 30.0

2. Secondary Outcome: Pharmacokinetics- 1)Plasma Concentration of TA-7284: Tmax,Cmax, AUC, Etc.; and 2)Urinary Excretion of TA-7284: Ae, Ae%, CLr
Time Frame: 19 days
Reporting Status: Not Posted

3. Secondary Outcome: Pharmacodynamics- 1)Urinary Glucose Excretion; 2)Plasma Glucose Concentration; 3)Insulin Concentration in Serum; 4)Insulinogenic Index;and 5)Hemoglobin A1c and Glycoalbumin
Time Frame: 18 days
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 19 days
Arm/Group | TA-7284 25 mg | TA-7284 100 mg | TA-7284 200 mg | TA-7284 400 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12 | 0/14 | 0/13 | 0/10
Other Adverse Events (participants affected / at risk) | 9/12 | 8/12 | 5/14 | 6/13 | 8/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TA-7284 25 mg (N=12) | TA-7284 100 mg (N=12) | TA-7284 200 mg (N=14) | TA-7284 400 mg (N=13) | Placebo (N=10)
Anaemia (Blood and lymphatic system disorders) | 0 | 2 | 1 | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 4 | 1 | 0 | 0 | 2
Stomatitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Toothache (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 1
Chills (General disorders) | 0 | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 1 | 0 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 0 | 1 | 0 | 0 | 3
Arthropod sting (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 2 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Syncope vasovagal (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Albumin urine present (Investigations) | 0 | 0 | 0 | 0 | 1
Beta 2 microglobulin urine increased (Investigations) | 0 | 0 | 1 | 0 | 0
Blood uric acid increased (Investigations) | 0 | 0 | 0 | 1 | 0
C-reactive protein increased (Investigations) | 0 | 0 | 0 | 1 | 0
Blood urine present (Investigations) | 0 | 0 | 0 | 1 | 0
N-telopeptide urine increased (Investigations) | 1 | 0 | 0 | 0 | 0
Urine ketone body present (Investigations) | 0 | 0 | 2 | 1 | 0
Fecal occult blood positive (Investigations) | 5 | 4 | 2 | 1 | 3
Deoxypyridinoline urine increased (Investigations) | 1 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other